CLINICAL TRIAL: NCT03594110
Title: A Multicentre International Randomized Parallel Group Double-blind Placebo-controlled Clinical Trial of EMPAgliflozin Once Daily to Assess Cardio-renal Outcomes in Patients With Chronic KIDNEY Disease
Brief Title: EMPA-KIDNEY (The Study of Heart and Kidney Protection With Empagliflozin)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: University of Oxford (Other); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245-0137; 2017-002971-24 (EudraCT Number)
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Empagliflozin 10 mg (Experimental): Patients with evidence of chronic kidney disease (CKD) at risk of kidney disease progression, with or without diagnosed diabetes mellitus administered orally once daily 10 milligram (mg) film-coated tablets of empagliflozin.
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator): Patients with evidence of chronic kidney disease (CKD) at risk of kidney disease progression, with or without diagnosed diabetes mellitus administered orally once daily film-coated tablets of placebo to match empagliflozin.
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Empagliflozin — Taken daily with or without food
  Arms: Empagliflozin 10 mg
Drug: Matching placebo — Taken daily with or without food
  Arms: Placebo

SUMMARY:
The primary aim of the study is to investigate the effect of empagliflozin on kidney disease progression or cardiovascular death versus placebo on top of standard of care in patients with pre-existing chronic kidney disease. After completion of the interventional part of the study (primary study completion) a subset of participants will be followed up in a post-trial observational (non-interventional) manner for cardio-renal outcomes (estimated study completion date).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years or at "full age" as required by local regulation
* Evidence of chronic kidney disease at risk of kidney disease progression defined by at least 3 months before and at the time of Screening Visit

  * CKD-EPI eGFR ≥20 to <45 mL/min/1.73m² or
  * CKD-EPI eGFR ≥45 to <90 mL/min/1.73m² with urinary albumin:creatinine ratio ≥200 mg/g (or protein:creatinine ratio ≥300 mg/g);
* Clinically appropriate doses of single agent RAS-inhibition with either ACEi or ARB unless such treatment is either not tolerated or not indicated
* A local Investigator judges that the participant neither requires empagliflozin (or any other SGLT-2 or SGLT-1/2 inhibitor), nor that such treatment is inappropriate;

Key Exclusion Criteria:

* Currently receiving SGLT-2 or SGLT-1/2 inhibitor
* Diabetes mellitus type 2 and prior atherosclerotic cardiovascular disease with an eGFR >60 mL/min/1.73m2 at Screening
* Receiving combined ACEi and ARB treatment
* Maintenance dialysis, functioning kidney transplant, or scheduled living donor transplant
* Polycystic kidney disease
* Previous or scheduled bariatric surgery
* Ketoacidosis in the past 5 years
* Symptomatic hypotension, or systolic blood pressure <90 or >180 mmHg at Screening
* ALT or AST >3x ULN at Screening
* Hypersensitivity to empagliflozin or other SGLT-2 inhibitor
* Any intravenous immunosuppression therapy in last 3 months; or anyone currently on >45 mg prednisolone (or equivalent)
* Use of an investigational medicinal product in the 30 days prior to Screening visit
* Known to be poorly compliant with clinic visits or prescribed medication
* Medical history that might limit the individual's ability to take trial treatments for the duration of the study (e.g. severe respiratory disease; history of cancer or evidence of spread within last 4 years, other than non-melanoma skin cancer; or recent history of alcohol or substance misuse)
* Current pregnancy, lactation or women of childbearing potential (WOCBP), unless using highly-effective contraception
* Type 1 diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6609 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2024-07-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (239):
- United States (47):
  - Nephrology Consultants, LLC, Huntsville, Alabama
  - Aventiv Research, Inc, Mesa, Arizona
  - Southern California Permanente Medical Group, San Diego, California
  - University of California Los Angeles, Sylmar, California
  - University of California Los Angeles, Torrance, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Chase Medical Research, LLC, Thomaston, Connecticut
  - Midland Florida Clinical Reearch Center, LLC, DeLand, Florida
  - University of Florida, Gainesville, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - East Coast Clinical Research, Inc, Lake City, Florida
  - Total Research Group, LLC, Miami, Florida
  - Hanson Clinical Research Center, Inc., Port Charlotte, Florida
  - Emory University, Atlanta, Georgia
  - The Jones Center for Diabetes and Endocrine Wellness, Macon, Georgia
  - Cedar Crosse Research Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Saint Elizabeth Healthcare, Covington, Kentucky
  - Lexington VA Health Care System - Troy Bowling Campus, Lexington, Kentucky
  - Medstar Health Research Institute, Baltimore, Maryland
  - Kidney Care and Transplant Services of New England, PC, West Springfield, Massachusetts
  - Saint Clair Specialty Physicians, Roseville, Michigan
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - VA Southern Nevada Healthcare System, North Las Vegas, Nevada
  - Seacoast Kidney and Hypertension Specialists, Portsmouth, New Hampshire
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Mountain Kidney and Hypertension Associates, PA, Asheville, North Carolina
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Brookview Hills Research Associates LLC, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Carolina Diabetes & Kidney Center, Sumter, South Carolina
  - Regional Health Clinical Research, Rapid City, South Dakota
  - Research Institute of Dallas, Dallas, Texas
  - Renal Disease Research Institute, Dallas, Texas
  - Academy Of Diabetes, Thyroid And Endocrine, PA, El Paso, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - P&I Clinical Research, LLC, Lufkin, Texas
  - Texas Institute for Kidney and Endocrine Disorders, Lufkin, Texas
  - Clinical Advancement Center PLLC, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Salem VA Medical Center, Salem, Virginia
  - Providence Medical Research Center, Spokane, Washington
- Canada (20):
  - Kelowna General Hospital, Kelowna, British Columbia
  - Kidney Care Centre - Surrey, Surrey, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - LMC Clinical Research Inc. (Brampton), Brampton, Ontario
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - LMC Clinical Research Inc. (Thornhill), Concord, Ontario
  - LMC Endocrinology Centres (Etobicoke) Ltd., Etobicoke, Ontario
  - London Health Science Centre, University Campus, London, Ontario
  - LMC Clinical Research Inc. (Ottawa), Nepean, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - LMC Clinical Research Inc. (Bayview), Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Fadia El Boreky Medicine Professional, Waterloo, Ontario
  - Clinical Research Solutions Inc., Waterloo, Ontario
  - Montreal Clinical Research Institute (IRCM), Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - CHUS Hopital Fleurimont, Sherbrooke, Quebec
  - CHU de Quebec-Universite Laval Research Centre, Québec
  - IUCPQ (Laval University), Québec
- China (16):
  - Beijing AnZhen Hospital, Beijing
  - Cardiovascular Institute and Fu Wai Hospital, Beijing
  - Xiangya Hospital, Central South University, Changsha
  - Xinqiao Hospital, Chongqing
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Jinzhou Central Hospital, Jinzhou
  - Jinling Hospital, Nanjing
  - Shanghai Fifth People's Hospital affiliated to Fudan University, Shanghai
  - Shenzhen People's Hospital, Shenzhen
  - Huazhong University of Science and Technology Union Shenzhen Hospital, Shenzhen
  - People's Hospital of Sichuan Province, Sichuan
  - SuZhou Kowloon Hospital, Suzhou
  - The Central Hospital of Wuhan, Wuhan
  - Wuhan Fourth Hospital, Wuhan
  - Henan Provincial People's Hospital, Zhengzhou
  - Zhuzhou Central Hospital, Zhuzhou
- Germany (36):
  - Studienzentrum Aschaffenburg, Aschaffenburg
  - Universitätsklinikum Augsburg, Augsburg
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen, Bad Oeynhausen
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Ärztezentrum Helle Mitte, Berlin
  - Klinikum Bielefeld gGmbH, Bielefeld
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Agaplesion Markus Krankenhaus, Frankfurt
  - ClinPhenomics GmbH & Co KG, Frankfurt, Frankfurt
  - Nierenzentrum Freiburg, Freiburg im Breisgau
  - Nephrologisches Zentrum Göttingen, Göttingen
  - Universitätsklinikum Halle/S., Halle
  - Zentrum für Nieren-, Hochdruck und Stoffwechselerkrankungen, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Dialysezentrum Heilbronn ÜBAG für Nephrologie und Dialyse, Heilbronn
  - Nephrologisches Zentrum Hoyerswerda, Hoyerswerda
  - Universitätsklinikum Jena, Jena
  - Städt. Klinikum, Karlsruhe, Moltkestr., Karlsruhe
  - Klinikum St. Georg gGmbH, Leipzig
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Mannheim GmbH, Mannheim
  - Nephrologisches Zentrum Mettmann, Mettmann
  - Klinikum der Universität München - Campus Innenstadt, München
  - Dialysezentrum Neckarsulm, Neckarsulm
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V., Nuremberg
  - MVZ Diaverum Potsdam, Potsdam
  - Universitätsklinikum Regensburg, Regensburg
  - Robert-Bosch-Krankenhaus GmbH, Stuttgart
  - Universitätsklinikum Ulm, Ulm
  - Nephrologisches Zentrum Velbert, Velbert
  - MVZ DaVita Viersen GmbH, Viersen
  - Nephrologisches Zentrum Villingen-Schwenningen, Villingen-Schwenningen
  - Gemeinschaftspraxis für Nephrologie und Rheumatologie, Wiesbaden
  - Universitätsklinikum Würzburg AÖR, Würzburg
- Italy (21):
  - Azienda Ospedaliera Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - A.O. Policlinico Giovanni XXIII di Bari, Bari
  - Policlinico S. Orsola Malpighi, Bologna
  - ASST degli Spedali Civili di Brescia, Brescia
  - A. O. Ospedale Civile di Vimercate e Circolo di Desio, Desio
  - Osp. S. Giovanni di Dio, Florence
  - Ospedale S. Cuore di Gesù, Gallipoli
  - Azienda Ospedaliera San Martino, Genova
  - Ospedale della Versilia, LIDO DI Camaiore (LU)
  - A.O.U.Policlinico G.Martino, Messina
  - Milano Fondazione IRCCS Ca'Granda-Ospedale Maggiore Policlinico, Milan
  - IRCCS San Raffaele, Milan
  - AOU Università degli Studi della Campania Luigi Vanvitelli, Napoli
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - A.O. Univ. Policlinico "Paolo Giaccone", Palermo
  - Poli Univ A. Gemelli, Roma
  - Azienda Ospedaliera Sant'Andrea-Università di Roma La Sapienza, Roma
  - IRCCS Ospedale "Casa Sollievo della Sofferenza", SAN Giovanni Rotondo (FG)
  - Ospedale Ignazio Veris delli Ponti, Scorrano (LE)
  - Ospedale Martini, Torino
  - A.O. Univ. Integrata di Verona, Verona
- Japan (25):
  - Aichi Medical University Hospital, Aichi
  - Chubu Rosai Hospital, Aichi, Nagoya
  - Fukui Prefectural Hospital, Fukui
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Joumou Ohashi Clinic, Gumma, Maebashi
  - Maebashi Hirosegawa Clinic, Gunma
  - Ota Diabetes Clinic, Gunma
  - University of Tsukuba Hospital, Ibaraki, Tsukuba
  - Medical Corporation Seijinkai Ikeda Hospital, Kagoshima
  - Tokai University Hospital, Kanagawa
  - Koukan Clinic, Kawasaki
  - Kobe University Hospital, Kobe
  - Tohoku University Hospital, Miyagi, Sendai
  - Nagoya University Hospital, Nagoya
  - Kawasaki Medical School Hospital, Okayama, Kurashiki
  - Okayama University Hospital, Okayama, Okayama
  - AMC Nishi-umeda Clinic, Osaka
  - Kansai Electric Power Hospital, Osaka
  - Iwasaki Internal Medicine Clinic, Osaka
  - Shiga University of Medical Science Hospital, Shiga, Otsu
  - Tokyo-Eki Center-building Clinic, Tokyo
  - Juntendo University Hospital, Tokyo, Bunkyo-ku
  - The University of Tokyo Hospital, Tokyo, Bunkyo-ku
  - Shin Clinic, Tokyo, Ota-ku
  - Center Hospital of the National Center for Global Health and Medicine, Tokyo, Shinjuku-ku
- Malaysia (21):
  - Hospital Sultanah Bahiyah, Alor Setar, Kedah
  - Hospital Ampang, Ampang
  - University Kebangsaan Malaysia, Cheras, Kuala Lumpur
  - Hospital Pulau Pinang, Georgetown, Pulau Pinang
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Sultanah Aminah, Johor Bahru
  - Hospital Kajang, Kajang, Selangor
  - Hospital Serdang, Kajang, Selangor
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University of Malaya Medical Centre, Kuala Lumpur
  - Hospital Selayang, Kuala Selangor
  - Hospital Sultanah Nur Zahirah, Kuala Terengganu
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Sarawak General Hospital, Kuching, Sarawak
  - Hospital Kulim, Kulim, Kedah
  - Hospital Melaka, Malacca
  - Hospital Pakar Sultanah Fatimah, Muar town
  - Hospital Tuanku Ja'afar, Seremban, Negeri Sembilan
  - Pusat Perubatan UiTM Jalan Hospital, Sungai Buloh
  - Hospital Sultan Abdul Halim, Sungai Petani
  - Hospital Taiping, Taiping, Perak
- United Kingdom (53):
  - Antrim Area Hospital, Antrim
  - Ulster Hospital, Belfast
  - Belfast City Hospital, Belfast
  - Queen Elizabeth Hospital, Birmingham
  - Oakenhurst Medical Practice, Blackburn
  - Royal Sussex County Hospital, Brighton
  - Southmead Hospital, Bristol
  - West Suffolk Hospital, Bury St Edmunds
  - Kent & Canterbury Hospital, Oncology Department, Canterbury, Canterbury
  - University Hospital of Wales, Cardiff
  - St Helier Hospital, Carshalton
  - Cheltenham General Hospital, Cheltenham
  - Hathaway Medical Centre, Chippenham
  - University Hospital Coventry, Coventry
  - Darent Valley Hospital, Chemotherapy Unit, Dartford
  - Royal Derby Hospital, Derby
  - Dorset County Hospital, Dorchester
  - Ninewells Hospital & Medical School, Dundee
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - Queen Elizabeth University Hospital, Glasgow
  - Gloucestershire Royal Hospital, Gloucester
  - Hull Royal Infirmary, Hull
  - Ipswich Hospital, Ipswich
  - Queen Elizabeth Hospital, Kings Lynn
  - St James's University Hospital, Leeds
  - University Hospitals of Leicester, Leicester
  - Aintree University Hospital, Liverpool
  - The Royal London Hospital, London
  - North Middlesex Hospital, London
  - Royal Free Hospital, London
  - King's College Hospital, London
  - St George's Hospital, London
  - Hammersmith Hospital, London
  - Altnagelvin Area Hospital, Londonderry
  - Freeman Hospital, Newcastle
  - Daisy Hill Hospital, Newry
  - Norfolk and Norwich University Hospital, Norwich
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - St Bartholomew's Medical Centre (OxFed), Oxford
  - Derriford Hospital, Plymouth
  - Wessex Kidney Centre, Portsmouth
  - Royal Berkshire Hospital, Reading
  - Queen's Hospital, Romford
  - Salford Royal Hospital, Salford
  - Northern General Hospital, Sheffield
  - Lister Hospital, Stevenage
  - University Hospitals of North Midlands, Stoke-on-Trent
  - Great Western Hospital, Swindon
  - Princess Royal Hospital, Telford
  - Royal Cornwall Hospital, Truro
  - Walsall Manor Hospital, Walsall

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website. The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Mottl A, Scott C, Green JB, Heerspink HJL, Mann JFE, McGill JB, Nangaku M, Rosenstock J, Rossing P, Li L, Li N, Vaduganathan M, Agarwal R; CONFIDENCE Trial Investigators. Baseline Kidney Function, Albuminuria, and Urine Albumin-Creatinine Ratio Reduction with Finerenone, Empagliflozin, or Both: Post Hoc Analyses of CONFIDENCE Trial. J Am Soc Nephrol. 2025 Nov 6. doi: 10.1681/ASN.0000000928. Online ahead of print. No abstract available. PMID 41196655
- [Derived] Uster A, Desai N, Navaneethan SD, Pfarr E, Mazo AR. Empagliflozin Reduces Risk of Hospitalization in Patients With Chronic Kidney Disease in the EMPA-KIDNEY Trial. Clin Ther. 2025 Dec;47(12):1091-1096. doi: 10.1016/j.clinthera.2025.09.005. Epub 2025 Oct 4. PMID 41047325
- [Derived] Zhou J, Williams C, Staplin N, Judge PK, Mayne KJ, Agrawal N, Arimoto R, Green JB, Cherney DZI, Tuttle KR, Leal J, Clarke P, Emberson JR, Preiss D, Wanner C, Landray MJ, Baigent C, Haynes R, Herrington WG, Mihaylova B; EMPA-KIDNEY Collaborative Group. Effects of empagliflozin on quality of life and healthcare use and costs in chronic kidney disease: a health economic analysis of the EMPA-KIDNEY trial. EClinicalMedicine. 2025 Jul 8;85:103338. doi: 10.1016/j.eclinm.2025.103338. eCollection 2025 Jul. PMID 40686671
- [Derived] Oshima M, Buizen L, Jongs N, Levin A, Chertow GM, Wheeler DC, Heerspink HJL, Arnott C, Jardine MJ, Mahaffey KW, Pollock C, Herrington WG, Perkovic V, Neuen BL. Sodium-Glucose Cotransporter 2 Inhibition and Hospitalizations in Patients with CKD: A Meta-Analysis of Kidney Outcome Trials. Clin J Am Soc Nephrol. 2025 Jul 14;20(9):1206-1214. doi: 10.2215/CJN.0000000771. PMID 40658498
- [Derived] Mayne KJ, Sardell RJ, Staplin N, Judge PK, Zhu D, Sammons E, Cherney DZI, Cheung AK, Maggioni AP, Nangaku M, Rossello X, Tuttle KR, Ihara K, Iwata T, Wanner C, Emberson J, Preiss D, Landray MJ, Baigent C, Haynes R, Herrington WG; EMPA-KIDNEY Collaborative Group. Frailty, Multimorbidity, and Polypharmacy: Exploratory Analyses of the Effects of Empagliflozin from the EMPA-KIDNEY Trial. Clin J Am Soc Nephrol. 2024 Sep 1;19(9):1119-1129. doi: 10.2215/CJN.0000000000000498. Epub 2024 Jun 27. PMID 40179340
- [Derived] EMPA-KIDNEY Collaborative Group; Herrington WG, Staplin N, Agrawal N, Wanner C, Green JB, Hauske SJ, Emberson JR, Preiss D, Judge P, Zhu D, Dayanandan R, Arimoto R, Mayne KJ, Ng SYA, Sammons E, Hill M, Stevens W, Wallendszus K, Brenner S, Cheung AK, Liu ZH, Li J, Hooi LS, Liu W, Kadowaki T, Nangaku M, Levin A, Cherney DZI, Maggioni AP, Pontremoli R, Deo R, Goto S, Rossello X, Tuttle KR, Steubl D, Massey D, Brueckmann M, Landray MJ, Baigent C, Haynes R; EMPA-KIDNEY Collaborative Group. Long-Term Effects of Empagliflozin in Patients with Chronic Kidney Disease. N Engl J Med. 2025 Feb 20;392(8):777-787. doi: 10.1056/NEJMoa2409183. Epub 2024 Oct 25. PMID 39453837
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Mayne KJ, Staplin N, Keane DF, Wanner C, Brenner S, Cejka V, Stegbauer J, Judge PK, Preiss D, Emberson J, Trinca D, Dayanandan R, Lee R, Nolan J, Omata A, Green JB, Cherney DZI, Hooi LS, Pontremoli R, Tuttle KR, Lees JS, Mark PB, Davies SJ, Hauske SJ, Steubl D, Bruckmann M, Landray MJ, Baigent C, Haynes R, Herrington WG; EMPA-KIDNEY Collaborative Group. Effects of Empagliflozin on Fluid Overload, Weight, and Blood Pressure in CKD. J Am Soc Nephrol. 2024 Feb 1;35(2):202-215. doi: 10.1681/ASN.0000000000000271. Epub 2023 Dec 12. PMID 38082486
- [Derived] EMPA-KIDNEY Collaborative Group. Impact of primary kidney disease on the effects of empagliflozin in patients with chronic kidney disease: secondary analyses of the EMPA-KIDNEY trial. Lancet Diabetes Endocrinol. 2024 Jan;12(1):51-60. doi: 10.1016/S2213-8587(23)00322-4. Epub 2023 Dec 4. PMID 38061372
- [Derived] EMPA-KIDNEY Collaborative Group. Effects of empagliflozin on progression of chronic kidney disease: a prespecified secondary analysis from the empa-kidney trial. Lancet Diabetes Endocrinol. 2024 Jan;12(1):39-50. doi: 10.1016/S2213-8587(23)00321-2. Epub 2023 Dec 4. PMID 38061371
- [Derived] The EMPA-KIDNEY Collaborative Group; Herrington WG, Staplin N, Wanner C, Green JB, Hauske SJ, Emberson JR, Preiss D, Judge P, Mayne KJ, Ng SYA, Sammons E, Zhu D, Hill M, Stevens W, Wallendszus K, Brenner S, Cheung AK, Liu ZH, Li J, Hooi LS, Liu W, Kadowaki T, Nangaku M, Levin A, Cherney D, Maggioni AP, Pontremoli R, Deo R, Goto S, Rossello X, Tuttle KR, Steubl D, Petrini M, Massey D, Eilbracht J, Brueckmann M, Landray MJ, Baigent C, Haynes R. Empagliflozin in Patients with Chronic Kidney Disease. N Engl J Med. 2023 Jan 12;388(2):117-127. doi: 10.1056/NEJMoa2204233. Epub 2022 Nov 4. PMID 36331190
- [Derived] Tuttle KR, Levin A, Nangaku M, Kadowaki T, Agarwal R, Hauske SJ, Elsasser A, Ritter I, Steubl D, Wanner C, Wheeler DC. Safety of Empagliflozin in Patients With Type 2 Diabetes and Chronic Kidney Disease: Pooled Analysis of Placebo-Controlled Clinical Trials. Diabetes Care. 2022 Jun 2;45(6):1445-1452. doi: 10.2337/dc21-2034. PMID 35472672
- [Derived] Almaimani M, Sridhar VS, Cherney DZI. Sodium-glucose cotransporter 2 inhibition in non-diabetic kidney disease. Curr Opin Nephrol Hypertens. 2021 Sep 1;30(5):474-481. doi: 10.1097/MNH.0000000000000724. PMID 34074889
- [Derived] Piperidou A, Loutradis C, Sarafidis P. SGLT-2 inhibitors and nephroprotection: current evidence and future perspectives. J Hum Hypertens. 2021 Jan;35(1):12-25. doi: 10.1038/s41371-020-00393-4. Epub 2020 Aug 10. PMID 32778748
- [Derived] Gonzalez DE, Foresto RD, Ribeiro AB. SGLT-2 inhibitors in diabetes: a focus on renoprotection. Rev Assoc Med Bras (1992). 2020 Jan 13;66Suppl 1(Suppl 1):s17-s24. doi: 10.1590/1806-9282.66.S1.17. PMID 31939531
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial with a interventional and a non-interventional part (post-trial follow-up). Interventional part: event-driven (ca. 1070 primary outcome events). Alongside the trial, a fraction of patients randomized in the interventional part gave consent to two sub-studies: body composition measurement and magnetic resonance imaging. Non-interventional part: patients who gave consent were observed for ca. 2 years.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Interventional Part
Arm/Group | Placebo | Empagliflozin 10 mg
Started | 3305 | 3304
Treated | 3305 | 3304
Body Composition Measurement (BCM) Sub-study (Patients included in the BCM sub-study) | 328 | 332
Magnetic Resonance Imaging (MRI) Sub-study (Patients included in the MRI sub-study) | 79 | 93
Completed (Patients who did not prematurely discontinue study treatment.) | 2457 | 2549
Not Completed | 848 | 755
Not completed — Participant concerned about study treatment | 23 | 28
Not completed — Doctor advice | 38 | 40
Not completed — Participants' wish | 89 | 68
Not completed — Adverse event-non-fatal events | 119 | 116
Not completed — Study drug stopped, reason missing | 336 | 294
Not completed — Cannot attend clinic because of personal problems | 8 | 16
Not completed — Cannot attend clinic because moving out of the area | 15 | 9
Not completed — Contraindicated drug started | 32 | 18
Not completed — Other reasons (include any category with a frequency <20 patients in total) | 58 | 45
Not completed — Adverse event-Serious fatal events | 130 | 121
Period: Non-interventional Part
Arm/Group | Placebo | Empagliflozin 10 mg
Started | 2419 (Patients entering the post-trial follow-up part) | 2472 (Patients entering the post-trial follow-up part)
Completed | 2371 | 2427
Not Completed | 48 | 45
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lost to Follow-up | 45 | 41

BASELINE CHARACTERISTICS:
Population: Randomised set (RS) included all randomised participants, whether treated or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Empagliflozin 10 mg | Total
Number analyzed (Participants) | 3305 | 3304 | 6609
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (13.9) | 63.4 (13.9) | 63.3 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1095 | 1097 | 2192
  Male | 2210 | 2207 | 4417
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 119 | 103 | 222
  Not Hispanic or Latino | 723 | 708 | 1431
  Unknown or Not Reported | 2463 | 2493 | 4956
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1920 | 1939 | 3859
  Black/ African-American | 134 | 128 | 262
  Asian | 1199 | 1194 | 2393
  Other including mixed race | 52 | 43 | 95

OUTCOME MEASURES:

1. Primary Outcome: Interventional Part: Time to First Occurrence of Kidney Disease Progression or Cardiovascular Death ('as Adjudicated')
Description: Time to first occurrence of kidney disease progression (KDP) or cardiovascular death is reported as incidence rate of first occurrence of KDP or adjudicated cardiovascular death.
  Incidence rate= (Number of patients who experienced the event of first occurrence of KDP or cardiovascular death)*100/(patient years at risk (pt-yrs at risk). pt-yrs at risk= sum of time at risk [days] over all patients in a treatment group / 365.25.
  Kidney disease progression was defined as:
  * end stage kidney disease (defined as the initiation of maintenance dialysis or receipt of a kidney transplant) OR
  * a sustained decline in estimated glomerular filtration rate (eGFR) to <10 mL/min/1.73m^2 OR
  * renal death OR
  * a sustained decline of ≥40% in eGFR from randomisation.
Time Frame: From the day of randomisation to the day of the final follow-up visit in the interventional part of the trial, up to 1136 days.
Population: Randomised set (RS) included all randomised participants, whether treated or not.
Measure: Number (95% Confidence Interval); unit: patients with events/100 pt-yrs at risk
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 3305 | 3304
patients with events/100 pt-yrs at risk | 8.96 [8.23 to 9.72] | 6.85 [6.22 to 7.51]
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Hazard ratio (HR) of the time to first occurrence of kidney disease progression or CV death. HR is based on a Cox regression model with terms for age, sex, screening diabetes status, local screening estimated glomerular filtration rate Chronic Kidney Disease Epidemiology Collaboration (eGFR (CKD-EPI)), local screening Urine albumin-to-creatinine ratio (UACR), region and treatment; Test type: Superiority — Null hypothesis: There is no difference between the effect of placebo and the effect of empagliflozin. Two-sided significance level of <0.0017 required at interim analysis; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.72, 99.83% CI 2-sided [0.59 to 0.89] — Comparison vs. Placebo

2. Secondary Outcome: Key Secondary Endpoint: Interventional Part - Time to First Hospitalization for Heart Failure ('as Adjudicated') or Cardiovascular Death ('as Adjudicated')
Description: Time to first hospitalization for heart failure ('as adjudicated') or cardiovascular death ('as adjudicated') is reported as incidence rate of first hospitalization for heart failure or cardiovascular death.
  Incidence rate= (Number of patients who experienced the event of first hospitalization for heart failure or cardiovascular death) *100/(patient years at risk (pt-yrs at risk)).
  pt-yrs at risk= sum of time at risk [days] over all patients in a treatment group / 365.25.
Time Frame: From the day of randomisation to the day of the final follow-up visit of the interventional part, up to 1140 days.
Population: Randomised set (RS) included all randomised participants, whether treated or not.
Measure: Number (95% Confidence Interval); unit: patients with events/100 pt-yrs at risk
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 3305 | 3304
patients with events/100 pt-yrs at risk | 2.39 [2.03 to 2.78] | 2.04 [1.70 to 2.40]
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Hazard ratio (HR) of the time to first hospitalization for heart failure or cardiovascular death. HR is based on a Cox regression model with terms for age, sex, screening diabetes status, local screening estimated glomerular filtration rate Chronic Kidney Disease Epidemiology Collaboration (eGFR (CKD-EPI)), local screening Urine albumin-to-creatinine ratio (UACR), region and treatment; Test type: Superiority — Null hypothesis: There is no difference between the effect of placebo and the effect of empagliflozin. Two-sided significance level of <0.0145 required at interim analysis; p = 0.1363, Regression, Cox; Hazard Ratio (HR) = 0.84, 98.55% CI 2-sided [0.63 to 1.12] — Comparison vs. Placebo

3. Secondary Outcome: Key Secondary Endpoint: Interventional Part - Time to Occurrences of All-cause Hospitalizations (First and Recurrent Combined)
Description: Time to occurrences of all-cause hospitalizations is reported as total number of all-cause hospitalizations (first and recurrent combined).
Time Frame: From the day of randomisation to the day of the final follow-up visit of the interventional part, up to 1140 days.
Population: Randomised set (RS) included all randomised participants, whether treated or not.
Measure: Number; unit: events (first and recurrent)
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 3305 | 3304
events (first and recurrent) | 1895 | 1612
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Hazard ratio (HR) of the time to occurrences of all-cause hospitalizations (first and recurrent combined). HR based on an analysis of recurrent events accounting for terminal events using a joint frailty model with terms for age, log(local screening UACR), local screening Chronic Kidney Disease Epidemiology Collaboration (eGFR (CKD-EPI)), treatment, sex, screening diabetes status, region; Test type: Superiority — Null hypothesis: There is no difference between the effect of placebo and the effect of empagliflozin. Two-sided significance level of <0.0097 required at interim analysis; p = 0.0022, Joint frailty model; Hazard Ratio (HR) = 0.86, 99.03% CI 2-sided [0.76 to 0.98] — Comparison vs. Placebo

4. Secondary Outcome: Key Secondary Endpoint: Interventional Part - Time to Death From Any Cause ('as Adjudicated')
Description: Time to death from any cause is reported as incidence rate of death from any cause.
  Incidence rate of death from any cause = (Number of patients who experienced the event of death from any cause) * 100/(patient years at risk (pt-yrs at risk)). pt-yrs at risk= sum of time at risk [days] over all patients in a treatment group / 365.25.
Time Frame: From the day of randomisation to the day of the final follow-up visit in the interventional part of the trial, up to 1140 days.
Population: Randomised set (RS) included all randomised participants, whether treated or not.
Measure: Number (95% Confidence Interval); unit: patients with events/100 pt-yrs at risk
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 3305 | 3304
patients with events/100 pt-yrs at risk | 2.59 [2.21 to 3.00] | 2.29 [1.94 to 2.68]
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Hazard ratio (HR) of the time to death from any cause. HR is based on a Cox regression model with terms for age, sex, screening diabetes status, local screening estimated glomerular filtration rate Chronic Kidney Disease Epidemiology Collaboration (eGFR (CKD-EPI)), local screening Urine albumin-to-creatinine ratio (UACR), region and treatment; Test type: Superiority — Null hypothesis: There is no difference between the effect of placebo and the effect of empagliflozin. Two-sided significance level of <0.0290 required at interim analysis; p = 0.2122, Regression, Cox; Hazard Ratio (HR) = 0.87, 97.1% CI 2-sided [0.68 to 1.11] — Comparison vs. Placebo

5. Secondary Outcome: Interventional Part: Time to First Occurrence of Kidney Disease Progression
Description: Time to first occurrence of kidney disease progression (KDP) is reported as incidence rate of first occurrence of kidney disease progression.
  Incidence rate of first occurrence of kidney disease progression= (Number of patients who experienced the event of first occurrence of kidney disease progression) *100/(patient years at risk (pt-yrs at risk)). pt-yrs at risk= sum of time at risk [days] over all patients in a treatment group / 365.25.
  Kidney disease progression was defined as:
  * end stage kidney disease (defined as the initiation of maintenance dialysis or receipt of a kidney transplant) OR
  * a sustained decline in estimated glomerular filtration rate (eGFR) to <10 mL/min/1.73m^2 OR
  * renal death OR
  * a sustained decline of ≥40% in eGFR from randomisation).
Time Frame: From the day of randomisation to the day of the final follow-up visit of the interventional part, up to 1136 days.
Population: Randomised set (RS) included all randomised participants, whether treated or not.
Measure: Number (95% Confidence Interval); unit: patients with events/100 pt-yrs at risk
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 3305 | 3304
patients with events/100 pt-yrs at risk | 8.09 [7.40 to 8.81] | 6.09 [5.50 to 6.72]
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Hazard ratio (HR) of the time to first occurrence of kidney disease progression. HR is based on a Cox regression model with terms for age, sex, screening diabetes status, local screening estimated glomerular filtration rate Chronic Kidney Disease Epidemiology Collaboration (eGFR (CKD-EPI)), local screening urine albumin-to-creatinine ratio (UACR), region and treatment; Test type: Superiority — Null hypothesis: There is no difference between the effect of placebo and the effect of empagliflozin; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.62 to 0.81] — Comparison vs. Placebo

6. Secondary Outcome: Interventional Part: Time to Cardiovascular Death ('as Adjudicated')
Description: Time to cardiovascular death ('as adjudicated') is reported as incidence rate of cardiovascular death.
  Incidence rate of cardiovascular death= (Number of patients who experienced the event of cardiovascular death) *100/(patient years at risk (pt-yrs at risk)). pt-yrs at risk= sum of time at risk [days] over all patients in a treatment group / 365.25.
Time Frame: From the day of randomisation to the day of the final follow-up visit of the interventional part, up to 1140 days.
Population: Randomised set (RS) included all randomised participants, whether treated or not.
Measure: Number (95% Confidence Interval); unit: patients with events/100 pt-yrs at risk
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 3305 | 3304
patients with events/100 pt-yrs at risk | 1.08 [0.84 to 1.35] | 0.91 [0.69 to 1.15]
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Hazard ratio (HR) of the time to cardiovascular death. HR is based on a Cox regression model with terms for age, sex, screening diabetes status, local screening estimated glomerular filtration rate Chronic Kidney Disease Epidemiology Collaboration (eGFR (CKD-EPI)), local screening urine albumin-to-creatinine ratio (UACR), region and treatment; Test type: Superiority — Null hypothesis: There is no difference between the effect of placebo and the effect of empagliflozin; p = 0.2932, Regression, Cox; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.59 to 1.17] — Comparison vs. Placebo

7. Secondary Outcome: Interventional Part: Time to First Occurrence Cardiovascular Death ('as Adjudicated') or End Stage Kidney Disease (ESKD)
Description: Time to first occurrence of cardiovascular death ('as adjudicated') or end stage kidney disease is reported as incidence rate of first occurrence of cardiovascular death or end stage kidney disease (ESKD).
  Incidence rate of first occurrence cardiovascular death or end stage kidney disease (ESKD)= (Number of patients who experienced the event of first occurrence of cardiovascular death or end stage kidney disease (ESKD)) *100/(patient years at risk (pt-yrs at risk)). pt-yrs at risk= sum of time at risk [days] over all patients in a treatment group / 365.25.
  ESKD was defined as the initiation of maintenance dialysis or receipt of a kidney transplant.
Time Frame: From the day of randomization to the day of the final follow-up visit in the interventional part of the trial, up to 1140 days.
Population: Randomised set (RS) included all randomised participants, whether treated or not.
Measure: Number (95% Confidence Interval); unit: patients with events/100 pt-yrs at risk
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 3305 | 3304
patients with events/100 pt-yrs at risk | 3.45 [3.01 to 3.92] | 2.55 [2.18 to 2.96]
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Hazard ratio (HR) of the time to first occurrence cardiovascular death or end stage kidney disease (ESKD). HR is based on a Cox regression model with terms for age, sex, screening diabetes status, local screening estimated glomerular filtration rate Chronic Kidney Disease Epidemiology Collaboration (eGFR (CKD-EPI)), local screening urine albumin-to-creatinine ratio (UACR), region and treatment; Test type: Superiority — Null hypothesis: There is no difference between the effect of placebo and the effect of empagliflozin; p = 0.0017, Regression, Cox; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.59 to 0.89] — Comparison vs. Placebo

8. Primary Outcome: Overall Study: Time to the First Occurrence of Kidney Disease Progression or Cardiovascular Death ('as Adjudicated')
Description: Time to first occurrence of kidney disease progression (KDP) or cardiovascular death is reported as incidence of progression of kidney disease or death from cardiovascular causes in the interventional part of the trial and in the post-trial follow-up (non-interventional part).
  Incidence rate= (Number of patients who experienced the event of first occurrence of KDP or cardiovascular death)*100/(patient years at risk (pt-yrs at risk). pt-yrs at risk= sum of time at risk [days] over all patients in a treatment group / 365.25.
  Kidney disease progression was defined as:
  * a sustained decline in eGFR to less than 10 mL/min/1.73m^2 OR
  * renal death OR
  * sustained decline of more than 40% in eGFR from randomization.
Time Frame: From the day of randomization in the interventional part of the trial until the individual day of end of study in the non-interventional part of the trial. Up to 1869 days.
Population: Randomised set (RS): included all randomised participants, whether treated or not.
Measure: Number (95% Confidence Interval); unit: patients with events/100 pt-yrs at risk
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 3305 | 3304
patients with events/100 pt-yrs at risk | 9.99 [9.38 to 10.62] | 8.36 [7.81 to 8.93]
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.72 to 0.87] — Comparison vs. Placebo

9. Secondary Outcome: Overall Study: Time to First Occurrence of Kidney Disease Progression
Description: The time to first occurrence of kidney disease progression in the interventional part of the trial and in the post-trial follow-up (non-interventional part) is reported as the incidence rate of first occurrence of kidney disease progression.
  Incidence rate of first occurrence of kidney disease progression= (Number of patients who experienced the event of first occurrence of kidney disease progression) *100/(patient years at risk (pt-yrs at risk)). pt-yrs at risk= sum of time at risk [days] over all patients in a treatment group / 365.25.
  Kidney disease progression was defined as:
  * end stage kidney disease (defined as the initiation of maintenance dialysis or receipt of a kidney transplant) OR
  * a sustained decline in estimated glomerular filtration rate (eGFR) to <10 mL/min/1.73m^2 OR
  * renal death OR
  * a sustained decline of ≥40% in eGFR from randomisation.
Time Frame: as for outcome 8
Population: Randomised set (RS) included all randomised participants, whether treated or not.
Measure: Number (95% Confidence Interval); unit: patients with events/100 pt-yrs at risk
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 3305 | 3304
patients with events/100 pt-yrs at risk | 8.95 [8.37 to 9.55] | 7.52 [7.00 to 8.06]
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; [analysis description as in outcome 5, analysis 1]; Test type: Other; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.72 to 0.87] — Comparison vs. Placebo

10. Secondary Outcome: Overall Study: Time to First Occurrence of Death From Any Cause or ESKD
Description: Time to first occurrence of death from any cause or end stage kidney disease (ESKD) in the interventional part of the trial and in the post-trial follow-up (non-interventional part) is reported as incidence rate of first occurrence of death from any cause or ESKD.
  Incidence rate of first occurrence of death from any cause or end stage kidney disease (ESKD)= (Number of patients who experienced the event of first occurrence of death any cause or end stage kidney disease (ESKD)) *100/(patient years at risk (pt-yrs at risk)). pt-yrs at risk= sum of time at risk [days] over all patients in a treatment group / 365.25.
  ESKD was defined as the initiation of maintenance dialysis or receipt of a kidney transplant.
Time Frame: as for outcome 8
Population: Randomised set (RS) included all randomised participants, whether treated or not.
Measure: Number (95% Confidence Interval); unit: patients with events/100 pt-yrs at risk
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 3305 | 3304
patients with events/100 pt-yrs at risk | 6.08 [5.62 to 6.55] | 5.13 [4.71 to 5.56]
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Hazard ratio (HR) of the time to first occurrence of death from any cause or ESKD. HR is based on a Cox regression model with terms for age, sex, screening diabetes status, local screening estimated glomerular filtration rate Chronic Kidney Disease Epidemiology Collaboration (eGFR (CKD-EPI)), local screening urine albumin-to-creatinine ratio (UACR), region and treatment; Test type: Other; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.72 to 0.90] — Comparison vs. Placebo

11. Secondary Outcome: Overall Study: Time to First Occurrence of ESKD
Description: Time to first occurrence of end stage kidney disease (ESKD) in the interventional part of the trial and in the post-trial follow-up (non-interventional part) is reported as incidence rate of first occurrence of ESKD.
  Incidence rate of first occurrence of end stage kidney disease (ESKD)= (Number of patients who experienced the event of first occurrence of ESKD) *100/(patient years at risk (pt-yrs at risk)). pt-yrs at risk= sum of time at risk [days] over all patients in a treatment group / 365.25.
  ESKD was defined as the initiation of maintenance dialysis or receipt of a kidney transplant.
Time Frame: as for outcome 8
Population: Randomised set (RS) included all randomised participants, whether treated or not.
Measure: Number (95% Confidence Interval); unit: patients with events/100 pt-yrs at risk
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 3305 | 3304
patients with events/100 pt-yrs at risk | 3.49 [3.14 to 3.85] | 2.72 [2.41 to 3.03]
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Hazard ratio (HR) of ESKD. HR is based on a Cox regression model with terms for age, sex, screening diabetes status, local screening estimated glomerular filtration rate Chronic Kidney Disease Epidemiology Collaboration (eGFR (CKD-EPI)), local screening urine albumin-to-creatinine ratio (UACR), region and treatment; Test type: Other; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.64 to 0.87] — Comparison vs. Placebo

12. Secondary Outcome: Body Composition Measurement Sub-study: Mean Absolute Fluid Overload, Averaged Over Time
Description: Mean absolute fluid overload averaged over time in the body composition measurement sub-study. Fluid overload or overhydration was measured using bioimpedance spectroscopy which derives the amount of water in liters (L) in the adipose tissue and lean mass tissues and computed as the difference between expected (based upon weight and body composition) versus measured extracellular water volume, with positive values representing excess fluid.
  A mixed model of repeated measures (MMRM) with terms for baseline, age, sex, screening diabetes status, local screening eGFR, local screening UACR, treatment, treatment-by-time interaction and baseline-by-time interaction was used for the analysis. The weighted mean of the values at 2 and 18 months.
Time Frame: MMRM included measurements at baseline, 2 months, and 18 months.
Population: Body composition measurement sub-study: all randomized patients who signed the informed consent form to participate in the body composition measurement sub-study, whether treated or not, with at least one valid BCM measurement. Patients with non-valid follow-up measurements were excluded from the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 309 | 311
Liters | 0.34 (0.05) | 0.10 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; A mixed model of repeated measures (MMRM) with terms for baseline, age, sex, screening diabetes status, local screening eGFR, local screening UACR, treatment, treatment-by-time interaction and baseline-by-time interaction; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.24, 95% CI 2-sided [-0.38 to -0.11] — [Comparator] - [Placebo]

13. Secondary Outcome: Magnetic Resonance Imaging Sub-study: Kidney Cortical T1 Mapping as Measured by Modified Look-Locker Inversion Recovery (MOLLI) at 18 Months
Description: Kidney cortical T1 mapping using the modified Look-Locker inversion recovery (MOLLI) measured by magnetic resonance imaging (MRI) in the placebo and empagliflozin groups.
  A linear regression with terms for age, sex, screening diabetes status, local screening eGFR, local screening UACR was used in the analysis.
Time Frame: At 18 months.
Population: Magnetic resonance imaging sub-study: all randomized patients who signed the informed consent form to participate in magnetic resonance imaging sub-study, whether treated or not.
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 79 | 93
milliseconds | 1634 (11) | 1622 (10)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Differences in MRI measurements between treatment groups were assessed using a linear regression with terms for age, sex, screening diabetes status, local screening eGFR, local screening UACR was used in the analysis; Test type: Other; p = 0.41, Regression, Linear; Mean Difference (Net) = -12, 95% CI 2-sided [-42 to 17] — [Comparator]-[Placebo]

ADVERSE EVENTS:
Time Frame: All-cause Mortality: From randomisation until end of study, up to 1869 days. Adverse events reporting: From randomisation until 7 days (Residual Effect Period) after the last drug intake, up to 1147 days.
Description: All-cause Mortality: Randomized set (RS): all randomized patients, whether treated or not.
  Adverse events reporting: Treated Set (TS): all patients who were dispensed randomized study medication.
  Only protocol pre-specified non-serious Adverse Events (AEs) were collected.
Arm/Group | Placebo | Empagliflozin 10 mg
All-Cause Mortality (participants affected / at risk) | 353/3305 | 314/3304
Serious Adverse Events (participants affected / at risk) | 1167/3305 | 1089/3304
Other Adverse Events (participants affected / at risk) | 262/3305 | 228/3304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3305) | Empagliflozin 10 mg (N=3304)
Anaemia (Blood and lymphatic system disorders) | 10 | 2
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 2
Aplasia pure red cell (Blood and lymphatic system disorders) | 1 | 0
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 2 | 2
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 5 | 6
Angina pectoris (Cardiac disorders) | 19 | 8
Angina unstable (Cardiac disorders) | 9 | 11
Aortic valve disease (Cardiac disorders) | 2 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 7 | 4
Arrhythmia (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 32 | 18
Atrial flutter (Cardiac disorders) | 4 | 4
Atrioventricular block (Cardiac disorders) | 2 | 3
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 2
Bradyarrhythmia (Cardiac disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 2 | 5
Bundle branch block (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 44 | 41
Cardiac fibrillation (Cardiac disorders) | 1 | 2
Cardiac sarcoidosis (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 14 | 7
Coronary artery stenosis (Cardiac disorders) | 4 | 3
Coronary vein stenosis (Cardiac disorders) | 1 | 0
Hypertensive cardiomyopathy (Cardiac disorders) | 10 | 5
Ischaemic cardiomyopathy (Cardiac disorders) | 45 | 33
Malignant hypertensive heart disease (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 3 | 0
Myocardial infarction (Cardiac disorders) | 31 | 39
Myocarditis (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 4 | 1
Pericardial effusion (Cardiac disorders) | 1 | 2
Pericarditis (Cardiac disorders) | 2 | 0
Pulseless electrical activity (Cardiac disorders) | 1 | 0
Sinus arrest (Cardiac disorders) | 1 | 1
Sinus bradycardia (Cardiac disorders) | 3 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 2 | 2
Trifascicular block (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 3
Ventricular extrasystoles (Cardiac disorders) | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 2 | 2
Ventricular tachyarrhythmia (Cardiac disorders) | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 2
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1 | 0
Congenital vesicoureteric reflux (Congenital, familial and genetic disorders) | 0 | 1
Heart block congenital (Congenital, familial and genetic disorders) | 0 | 1
Myocardial bridging (Congenital, familial and genetic disorders) | 1 | 0
Osteoporosis-pseudoglioma syndrome (Congenital, familial and genetic disorders) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 1 | 0
Thalassaemia (Congenital, familial and genetic disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 2 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 4
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0
Thyroiditis (Endocrine disorders) | 0 | 1
Amaurosis fugax (Eye disorders) | 2 | 1
Cataract (Eye disorders) | 3 | 3
Diabetic eye disease (Eye disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 2
Glaucoma (Eye disorders) | 1 | 0
Lacrimal disorder (Eye disorders) | 0 | 1
Lens dislocation (Eye disorders) | 1 | 0
Macular degeneration (Eye disorders) | 1 | 3
Retinal artery occlusion (Eye disorders) | 1 | 1
Retinal detachment (Eye disorders) | 2 | 2
Retinal haemorrhage (Eye disorders) | 1 | 0
Retinal tear (Eye disorders) | 2 | 0
Retinopathy proliferative (Eye disorders) | 0 | 1
Ulcerative keratitis (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 3
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 7
Anal fissure (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 1
Chronic gastrointestinal bleeding (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 3 | 2
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 3
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 4 | 1
Gastrointestinal fistula (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 6
Gastrointestinal ischaemia (Gastrointestinal disorders) | 2 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 3
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 2 | 0
Ileus paralytic (Gastrointestinal disorders) | 3 | 0
Inguinal hernia (Gastrointestinal disorders) | 4 | 3
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 4 | 1
Intestinal polyp (Gastrointestinal disorders) | 7 | 4
Jejunal perforation (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 5
Mechanical ileus (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 1 | 2
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 2 | 2
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0
Pancreatic mass (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 5 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Retroperitoneal fibrosis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Umbilical hernia (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 10 | 2
Varices oesophageal (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 4
Autoresuscitation (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 12 | 7
Death (General disorders) | 10 | 10
Gait disturbance (General disorders) | 3 | 0
General physical health deterioration (General disorders) | 3 | 0
Incarcerated hernia (General disorders) | 1 | 0
Necrosis (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 4
Oedema (General disorders) | 4 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 2 | 4
Sudden cardiac death (General disorders) | 17 | 12
Sudden death (General disorders) | 1 | 0
Vascular stent occlusion (General disorders) | 1 | 1
Vascular stent thrombosis (General disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 4
Cholecystitis (Hepatobiliary disorders) | 6 | 9
Cholelithiasis (Hepatobiliary disorders) | 2 | 6
Gallbladder necrosis (Hepatobiliary disorders) | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 4 | 3
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 2
Hepatitis cholestatic (Hepatobiliary disorders) | 2 | 1
Hepatitis toxic (Hepatobiliary disorders) | 4 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 7 | 5
Non-alcoholic fatty liver (Hepatobiliary disorders) | 2 | 2
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Allergy to vaccine (Immune system disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 1
Abdominal sepsis (Infections and infestations) | 1 | 2
Abscess (Infections and infestations) | 2 | 2
Abscess soft tissue (Infections and infestations) | 0 | 2
Appendicitis (Infections and infestations) | 1 | 5
Arthritis infective (Infections and infestations) | 1 | 2
Bacterial infection (Infections and infestations) | 2 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Bone abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 4 | 2
Bronchitis bacterial (Infections and infestations) | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1
Candida infection (Infections and infestations) | 0 | 1
Cardiac valve abscess (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 12 | 9
Cellulitis gangrenous (Infections and infestations) | 1 | 0
Clostridium colitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Corona virus infection (Infections and infestations) | 107 | 98
Cystitis (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 1 | 1
Diabetic foot infection (Infections and infestations) | 6 | 17
Diabetic gangrene (Infections and infestations) | 1 | 4
Diarrhoea infectious (Infections and infestations) | 1 | 2
Diverticulitis (Infections and infestations) | 6 | 7
Ear infection (Infections and infestations) | 1 | 1
Empyema (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 3 | 0
Endocarditis bacterial (Infections and infestations) | 3 | 0
Enterobacter sepsis (Infections and infestations) | 0 | 1
Epstein-Barr virus infection (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Gallbladder empyema (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 10 | 8
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Gastrointestinal bacterial infection (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 2 | 0
Genital infection fungal (Infections and infestations) | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 1
Helicobacter gastritis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 3 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 | 2
Influenza (Infections and infestations) | 1 | 1
Inguinal hernia gangrenous (Infections and infestations) | 0 | 1
Joint abscess (Infections and infestations) | 1 | 2
Labyrinthitis (Infections and infestations) | 1 | 0
Laryngitis bacterial (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 4
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 2
Lymphangitis (Infections and infestations) | 0 | 1
Meningoencephalitis bacterial (Infections and infestations) | 1 | 0
Muscle abscess (Infections and infestations) | 2 | 0
Nail infection (Infections and infestations) | 1 | 0
Necrotising soft tissue infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Oral infection (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 0 | 2
Osteomyelitis (Infections and infestations) | 1 | 3
Osteomyelitis acute (Infections and infestations) | 0 | 1
Osteomyelitis bacterial (Infections and infestations) | 1 | 1
Osteomyelitis chronic (Infections and infestations) | 1 | 2
Otitis externa (Infections and infestations) | 1 | 0
Pancreatic abscess (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 1
Peritonitis (Infections and infestations) | 1 | 1
Peritonitis bacterial (Infections and infestations) | 2 | 0
Pleural infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 42 | 39
Pneumonia bacterial (Infections and infestations) | 4 | 7
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 1
Prostate infection (Infections and infestations) | 1 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0
Psoas abscess (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 2 | 0
Pyelocystitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 3 | 3
Pyelonephritis acute (Infections and infestations) | 1 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Renal abscess (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 4 | 2
Respiratory tract infection viral (Infections and infestations) | 0 | 2
Retroperitoneal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 6 | 8
Septic shock (Infections and infestations) | 1 | 2
Severe invasive streptococcal infection (Infections and infestations) | 0 | 1
Skin bacterial infection (Infections and infestations) | 2 | 2
Skin infection (Infections and infestations) | 1 | 2
Soft tissue infection (Infections and infestations) | 0 | 1
Spinal cord abscess (Infections and infestations) | 1 | 1
Staphylococcal infection (Infections and infestations) | 1 | 2
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Streptococcal infection (Infections and infestations) | 0 | 2
Streptococcal sepsis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 2 | 1
Systemic bacterial infection (Infections and infestations) | 1 | 0
Thrombophlebitis septic (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 4
Upper respiratory tract infection bacterial (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 31 | 27
Urinary tract infection bacterial (Infections and infestations) | 6 | 7
Urosepsis (Infections and infestations) | 5 | 6
Viral diarrhoea (Infections and infestations) | 1 | 2
Viral infection (Infections and infestations) | 2 | 1
Viral pericarditis (Infections and infestations) | 1 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Wound abscess (Infections and infestations) | 0 | 2
Wound infection (Infections and infestations) | 1 | 2
Wound infection bacterial (Infections and infestations) | 0 | 1
Wound sepsis (Infections and infestations) | 0 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 3 | 6
Back injury (Injury, poisoning and procedural complications) | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 2
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 2
Concussion (Injury, poisoning and procedural complications) | 0 | 2
Coronary artery restenosis (Injury, poisoning and procedural complications) | 3 | 0
Crush injury (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 3 | 1
Fall (Injury, poisoning and procedural complications) | 19 | 17
Femoral neck fracture (Injury, poisoning and procedural complications) | 5 | 3
Femur fracture (Injury, poisoning and procedural complications) | 9 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 2 | 5
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 1
Foreign body aspiration (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 2
Fractured ischium (Injury, poisoning and procedural complications) | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 5
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 7 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 5
Inadequate haemodialysis (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 3
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Oesophageal injury (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 1
Post angioplasty restenosis (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 2
Rib fracture (Injury, poisoning and procedural complications) | 5 | 4
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 2
Skin injury (Injury, poisoning and procedural complications) | 1 | 2
Skin wound (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal cord injury lumbar (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 2
Splenic injury (Injury, poisoning and procedural complications) | 0 | 1
Stab wound (Injury, poisoning and procedural complications) | 0 | 2
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 3 | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Tendon injury (Injury, poisoning and procedural complications) | 2 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 3
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 2 | 3
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Vascular injury (Injury, poisoning and procedural complications) | 1 | 0
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2
Angiogram (Investigations) | 0 | 4
Angiogram peripheral (Investigations) | 1 | 2
Anticoagulation drug level above therapeutic (Investigations) | 0 | 1
Arteriogram carotid (Investigations) | 0 | 1
Arteriogram coronary (Investigations) | 2 | 3
Biopsy intestine (Investigations) | 0 | 2
Biopsy kidney (Investigations) | 3 | 6
Biopsy liver (Investigations) | 3 | 0
Biopsy prostate (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 56 | 43
Blood glucose increased (Investigations) | 3 | 0
Blood magnesium decreased (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 3 | 1
Blood potassium increased (Investigations) | 87 | 76
Blood pressure decreased (Investigations) | 4 | 4
Blood pressure increased (Investigations) | 1 | 1
Blood sodium decreased (Investigations) | 1 | 1
Bronchoscopy (Investigations) | 1 | 1
Catheterisation cardiac (Investigations) | 11 | 8
Colonoscopy (Investigations) | 9 | 1
Computerised tomogram (Investigations) | 0 | 1
Coronavirus test positive (Investigations) | 3 | 6
Cystoscopy (Investigations) | 1 | 0
Endoscopy gastrointestinal (Investigations) | 2 | 3
Endoscopy upper gastrointestinal tract (Investigations) | 1 | 2
Heart rate irregular (Investigations) | 1 | 1
Investigation (Investigations) | 2 | 4
Laryngoscopy (Investigations) | 0 | 1
Nuclear magnetic resonance imaging abdominal (Investigations) | 1 | 0
Sleep study (Investigations) | 1 | 1
Ultrasound kidney (Investigations) | 0 | 1
Ultrasound liver (Investigations) | 1 | 0
Ultrasound scan (Investigations) | 1 | 0
Ureteroscopy (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 20 | 22
Diabetes mellitus (Metabolism and nutrition disorders) | 23 | 19
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 6 | 5
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 5
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 9 | 4
Fluid retention (Metabolism and nutrition disorders) | 3 | 0
Gout (Metabolism and nutrition disorders) | 5 | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 14 | 8
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 4 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 14 | 14
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 11 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 3
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 4
Insulin-requiring type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Ketosis (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 6
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 9 | 8
Uraemic acidosis (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 2 | 3
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 3 | 1
Joint destruction (Musculoskeletal and connective tissue disorders) | 2 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 10 | 4
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 | 4
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 4 | 3
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Adenosquamous cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenosquamous cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 11
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 6
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer male (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoid tumour of the prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoma in situ of penis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Clear cell sarcoma of the kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ear neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Enchondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Follicle centre lymphoma, follicular grade I, II, III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2
Hepatic cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Osteosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Pancreatic carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Peritoneal sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Plasma cell myeloma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 8
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 6
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Thymoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transformation to acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal ganglia infarction (Nervous system disorders) | 0 | 1
Basilar artery thrombosis (Nervous system disorders) | 1 | 0
Brain stem infarction (Nervous system disorders) | 0 | 1
Carotid artery aneurysm (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 2 | 0
Cerebellar infarction (Nervous system disorders) | 2 | 1
Cerebral infarction (Nervous system disorders) | 3 | 2
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cranial nerve paralysis (Nervous system disorders) | 1 | 2
Dementia (Nervous system disorders) | 1 | 1
Dementia Alzheimer's type (Nervous system disorders) | 1 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 5 | 3
Dizziness postural (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 2 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 6 | 10
Headache (Nervous system disorders) | 2 | 6
Hemiplegia (Nervous system disorders) | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 0 | 1
Hypoglycaemic encephalopathy (Nervous system disorders) | 1 | 0
Hypoglycaemic unconsciousness (Nervous system disorders) | 2 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 34 | 30
Lacunar infarction (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 3 | 1
Microvascular cranial nerve palsy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Movement disorder (Nervous system disorders) | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 2
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 2
Post stroke seizure (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 6 | 0
Sciatica (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 2 | 4
Speech disorder (Nervous system disorders) | 0 | 1
Spinal cord herniation (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 8 | 16
Tension headache (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 14 | 12
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
Visual field defect (Nervous system disorders) | 1 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Acute psychosis (Psychiatric disorders) | 2 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Bipolar disorder (Psychiatric disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 3 | 2
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Mania (Psychiatric disorders) | 1 | 0
Psychotic behaviour (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 117 | 93
Calculus urethral (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 1
Diabetic end stage renal disease (Renal and urinary disorders) | 4 | 5
Diabetic nephropathy (Renal and urinary disorders) | 9 | 4
End stage renal disease (Renal and urinary disorders) | 27 | 35
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 | 1
Glomerulonephritis (Renal and urinary disorders) | 1 | 0
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 2 | 0
Glomerulonephritis membranous (Renal and urinary disorders) | 7 | 3
Haematuria (Renal and urinary disorders) | 0 | 3
Hydronephrosis (Renal and urinary disorders) | 1 | 4
IgA nephropathy (Renal and urinary disorders) | 5 | 4
Lupus nephritis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Nephrotic syndrome (Renal and urinary disorders) | 1 | 1
Oliguria (Renal and urinary disorders) | 0 | 1
Paraneoplastic nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 2 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 2 | 2
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 3 | 3
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 3
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1
Ovarian failure (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Combined pulmonary fibrosis and emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 6 | 3
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 2
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Social problem (Social circumstances) | 0 | 2
Aneurysm repair (Surgical and medical procedures) | 1 | 0
Angioplasty (Surgical and medical procedures) | 2 | 3
Ankle operation (Surgical and medical procedures) | 2 | 0
Aortic aneurysm repair (Surgical and medical procedures) | 4 | 1
Aortic valve repair (Surgical and medical procedures) | 0 | 1
Aortic valve replacement (Surgical and medical procedures) | 2 | 3
Appendicectomy (Surgical and medical procedures) | 3 | 2
Arterial bypass operation (Surgical and medical procedures) | 1 | 0
Arterial repair (Surgical and medical procedures) | 1 | 0
Arterial stent insertion (Surgical and medical procedures) | 2 | 2
Arteriovenous fistula operation (Surgical and medical procedures) | 8 | 4
Arteriovenous shunt operation (Surgical and medical procedures) | 12 | 8
Bladder catheter removal (Surgical and medical procedures) | 1 | 0
Bladder catheterisation (Surgical and medical procedures) | 0 | 2
Bladder lesion excision (Surgical and medical procedures) | 1 | 1
Bladder operation (Surgical and medical procedures) | 1 | 2
Bladder polypectomy (Surgical and medical procedures) | 1 | 0
Bone debridement (Surgical and medical procedures) | 0 | 3
Bone operation (Surgical and medical procedures) | 0 | 2
CSF shunt operation (Surgical and medical procedures) | 1 | 0
Cardiac ablation (Surgical and medical procedures) | 4 | 5
Cardiac operation (Surgical and medical procedures) | 2 | 0
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 1 | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 12 | 10
Cardiac pacemaker removal (Surgical and medical procedures) | 0 | 1
Cardiac pacemaker replacement (Surgical and medical procedures) | 3 | 4
Cardiac resynchronisation therapy (Surgical and medical procedures) | 1 | 0
Cardioversion (Surgical and medical procedures) | 1 | 3
Carotid artery stent insertion (Surgical and medical procedures) | 1 | 0
Carotid endarterectomy (Surgical and medical procedures) | 0 | 3
Cataract operation (Surgical and medical procedures) | 27 | 12
Chemotherapy (Surgical and medical procedures) | 1 | 1
Chest wall operation (Surgical and medical procedures) | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 7 | 5
Colectomy (Surgical and medical procedures) | 1 | 1
Colostomy (Surgical and medical procedures) | 0 | 1
Colostomy closure (Surgical and medical procedures) | 1 | 0
Coronary angioplasty (Surgical and medical procedures) | 2 | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 3 | 5
Coronary artery bypass (Surgical and medical procedures) | 8 | 1
Cyst removal (Surgical and medical procedures) | 0 | 2
Dialysis device insertion (Surgical and medical procedures) | 19 | 11
Ear operation (Surgical and medical procedures) | 0 | 1
Elbow operation (Surgical and medical procedures) | 1 | 1
Endarterectomy (Surgical and medical procedures) | 0 | 1
Endometrial ablation (Surgical and medical procedures) | 1 | 0
External fixation of fracture (Surgical and medical procedures) | 0 | 1
Eye operation (Surgical and medical procedures) | 1 | 2
Eyelid operation (Surgical and medical procedures) | 0 | 2
Foot amputation (Surgical and medical procedures) | 1 | 5
Fracture treatment (Surgical and medical procedures) | 2 | 2
Gallbladder operation (Surgical and medical procedures) | 1 | 2
Gastric operation (Surgical and medical procedures) | 1 | 1
Gastric stapling (Surgical and medical procedures) | 1 | 1
Gastrointestinal surgery (Surgical and medical procedures) | 1 | 0
Glaucoma surgery (Surgical and medical procedures) | 2 | 0
Haemorrhoid operation (Surgical and medical procedures) | 1 | 4
Heart valve replacement (Surgical and medical procedures) | 1 | 0
Hepatectomy (Surgical and medical procedures) | 1 | 0
Hepatic embolisation (Surgical and medical procedures) | 0 | 1
Hernia repair (Surgical and medical procedures) | 5 | 4
Hip arthroplasty (Surgical and medical procedures) | 4 | 3
Hip surgery (Surgical and medical procedures) | 6 | 6
Hospitalisation (Surgical and medical procedures) | 13 | 10
Hysterectomy (Surgical and medical procedures) | 2 | 3
Implantable defibrillator insertion (Surgical and medical procedures) | 1 | 3
Implantable defibrillator replacement (Surgical and medical procedures) | 3 | 3
Intervertebral disc operation (Surgical and medical procedures) | 2 | 4
Intestinal polypectomy (Surgical and medical procedures) | 6 | 5
Intra-cerebral aneurysm operation (Surgical and medical procedures) | 1 | 0
Joint arthroplasty (Surgical and medical procedures) | 3 | 0
Joint surgery (Surgical and medical procedures) | 2 | 1
Knee arthroplasty (Surgical and medical procedures) | 4 | 9
Knee operation (Surgical and medical procedures) | 10 | 6
Large intestine operation (Surgical and medical procedures) | 0 | 2
Leg amputation (Surgical and medical procedures) | 1 | 7
Liver operation (Surgical and medical procedures) | 0 | 1
Low density lipoprotein apheresis (Surgical and medical procedures) | 0 | 1
Lung operation (Surgical and medical procedures) | 2 | 0
Mastectomy (Surgical and medical procedures) | 3 | 0
Meniscus operation (Surgical and medical procedures) | 3 | 0
Middle ear operation (Surgical and medical procedures) | 0 | 1
Mitral valve repair (Surgical and medical procedures) | 2 | 0
Nasal operation (Surgical and medical procedures) | 0 | 2
Nephrectomy (Surgical and medical procedures) | 0 | 3
Oesophageal operation (Surgical and medical procedures) | 0 | 1
Oophorectomy (Surgical and medical procedures) | 2 | 0
Open reduction of fracture (Surgical and medical procedures) | 0 | 1
Oral surgery (Surgical and medical procedures) | 1 | 0
Ovarian operation (Surgical and medical procedures) | 1 | 0
Packed red blood cell transfusion (Surgical and medical procedures) | 0 | 2
Pain management (Surgical and medical procedures) | 2 | 1
Pancreatic operation (Surgical and medical procedures) | 0 | 1
Parathyroidectomy (Surgical and medical procedures) | 2 | 1
Pelvic floor repair (Surgical and medical procedures) | 1 | 0
Percutaneous coronary intervention (Surgical and medical procedures) | 3 | 0
Peripheral artery angioplasty (Surgical and medical procedures) | 7 | 3
Peripheral artery bypass (Surgical and medical procedures) | 1 | 3
Peripheral artery stent insertion (Surgical and medical procedures) | 4 | 5
Peripheral endarterectomy (Surgical and medical procedures) | 2 | 0
Peripheral revascularisation (Surgical and medical procedures) | 1 | 0
Prostatic operation (Surgical and medical procedures) | 1 | 2
Radical prostatectomy (Surgical and medical procedures) | 1 | 0
Radiotherapy (Surgical and medical procedures) | 3 | 0
Rectal prolapse repair (Surgical and medical procedures) | 1 | 0
Removal of foreign body from joint (Surgical and medical procedures) | 0 | 1
Removal of internal fixation (Surgical and medical procedures) | 1 | 1
Renal stone removal (Surgical and medical procedures) | 2 | 2
Retinal laser coagulation (Surgical and medical procedures) | 1 | 0
Retinal operation (Surgical and medical procedures) | 1 | 0
Shoulder operation (Surgical and medical procedures) | 5 | 0
Skin graft (Surgical and medical procedures) | 0 | 1
Spinal cord operation (Surgical and medical procedures) | 1 | 0
Spinal fusion surgery (Surgical and medical procedures) | 1 | 0
Spinal laminectomy (Surgical and medical procedures) | 0 | 2
Spinal operation (Surgical and medical procedures) | 5 | 2
Stem cell transplant (Surgical and medical procedures) | 0 | 1
Subdural haematoma evacuation (Surgical and medical procedures) | 0 | 1
Thoracic operation (Surgical and medical procedures) | 1 | 0
Thrombectomy (Surgical and medical procedures) | 1 | 0
Thyroid operation (Surgical and medical procedures) | 2 | 0
Thyroidectomy (Surgical and medical procedures) | 1 | 1
Toe amputation (Surgical and medical procedures) | 11 | 16
Tongue operation (Surgical and medical procedures) | 2 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 1
Tracheostomy (Surgical and medical procedures) | 1 | 0
Transmyocardial revascularisation (Surgical and medical procedures) | 1 | 0
Transurethral bladder resection (Surgical and medical procedures) | 2 | 1
Transurethral prostatectomy (Surgical and medical procedures) | 1 | 0
Tricuspid valve repair (Surgical and medical procedures) | 1 | 0
Ureteral stent insertion (Surgical and medical procedures) | 1 | 3
Ureteral stent removal (Surgical and medical procedures) | 0 | 2
Ureteric calculus removal (Surgical and medical procedures) | 0 | 1
Ureteric operation (Surgical and medical procedures) | 1 | 1
Uterine dilation and curettage (Surgical and medical procedures) | 1 | 1
Uterine operation (Surgical and medical procedures) | 1 | 0
Aortic aneurysm (Vascular disorders) | 3 | 3
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 1 | 1
Aortic dissection rupture (Vascular disorders) | 0 | 1
Aortic occlusion (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 1
Arterial stenosis (Vascular disorders) | 2 | 0
Blood pressure inadequately controlled (Vascular disorders) | 1 | 2
CT hypotension complex (Vascular disorders) | 1 | 1
Circulatory collapse (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 9 | 4
Haematoma (Vascular disorders) | 3 | 3
Hypertension (Vascular disorders) | 8 | 3
Hypertensive crisis (Vascular disorders) | 8 | 5
Hypertensive emergency (Vascular disorders) | 1 | 2
Hypovolaemic shock (Vascular disorders) | 1 | 1
Malignant hypertension (Vascular disorders) | 1 | 0
Necrosis ischaemic (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 2 | 0
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 1
Peripheral artery occlusion (Vascular disorders) | 2 | 1
Peripheral artery stenosis (Vascular disorders) | 2 | 1
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 2 | 1
Peripheral vascular disorder (Vascular disorders) | 2 | 4
Temporal arteritis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 2 | 4
Vein rupture (Vascular disorders) | 0 | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3305) | Empagliflozin 10 mg (N=3304)
Gout (Metabolism and nutrition disorders) | 262 | 228

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (8):
  • Study Protocol: EMPA-KIDNEY Clinical Trial Protocol (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/10/NCT03594110/Prot_000.pdf
  • Study Protocol: EMPA-KIDNEY Post-Trial Follow-Up Protocol (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT03594110/Prot_004.pdf
  • Study Protocol: EMPA-KIDNEY MRI Sub-study Protocol (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/10/NCT03594110/Prot_005.pdf
  • Study Protocol: EMPA-KIDNEY BCM Sub-study Protocol (2019-03-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT03594110/Prot_006.pdf
  • Statistical Analysis Plan: EMPA-KIDNEY: Trial Statistical Analysis Plan (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT03594110/SAP_001.pdf
  • Statistical Analysis Plan: EMPA-KIDNEY Post-Trial Follow-Up Data Analysis Plan (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT03594110/SAP_003.pdf
  • Statistical Analysis Plan: EMPA-KIDNEY BCM sub-study Data Analysis Plan (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT03594110/SAP_007.pdf
  • Statistical Analysis Plan: EMPA-KIDNEY MRI sub-study Data Analysis Plan (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT03594110/SAP_008.pdf